CLINICAL TRIAL: NCT02423603
Title: A Phase II, Double-blind, Randomised, Placebo-controlled Study of the AKT Inhibitor AZD5363 in Combination With Paclitaxel in Triple-Negative Advanced or Metastatic Breast Cancer (PAKT).
Brief Title: PAKT: AZD5363 in Combination With Paclitaxel in Triple-Negative Advanced or Metastatic Breast Cancer
Acronym: PAKT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 009246QM; 2013-001521-43 (EudraCT Number)
Record Dates: First submitted 2014-07-11; First posted 2015-04-22 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Triple Negative Breast Cancer; Metastatic; AKT Inhibitor; Advanced; AZD5363; Paclitaxel; PAKT; Capivasertib
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; capivasertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel + AZD5363 (Active Comparator): Paclitaxel was administered as a once-per-week intravenous infusion of 90 mg/m2 over approximately 1 hour on days 1, 8, and 15 of each 28-day treatment cycle. Capivasertib 400 mg was administered orally twice per day on an intermittent weekly dosing schedule, with treatment on days 2 to 5 of weeks 1, 2, and 3 within each 28-day cycle.
  Interventions: Drug: Paclitaxel; Drug: AZD5363
- Paclitaxel + Placebo (Placebo Comparator): Paclitaxel was administered as a once-per-week intravenous infusion of 90 mg/m2 over approximately 1 hour on days 1, 8, and 15 of each 28-day treatment cycle. Placebo was administered orally twice per day on an intermittent weekly dosing schedule, with treatment on days 2 to 5 of weeks 1, 2, and 3 within each 28-day cycle.
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Paclitaxel — Patient receive Once a week for three weeks - with one week off treatment
  Other Names: Taxol
Drug: AZD5363 — Patients receive AZD5363/Placebo in an intermittent treatment schedule. Please see study arms for full information.
  Other Names: Capivasertib
  Arms: Paclitaxel + AZD5363
Drug: Placebo — Patients receive AZD5363/Placebo in an intermittent treatment schedule. Please see study arms for full information.
  Arms: Paclitaxel + Placebo

SUMMARY:
PAKT was an investigator-led, placebo-controlled, randomized phase II trial performed in 42 academic medical centers in the United Kindom, South Korea, France, Hungary, Romania, and Georgia. Patients were randomly assigned (1:1) to receive paclitaxel plus capivasertib or paclitaxel plus placebo. Stratification was by number of metastatic sites (< 3 v ≥ 3) and interval from the end of prior adjuvant or neoadjuvant chemotherapy (≤ 12 v > 12 months v no prior chemotherapy).

Paclitaxel was administered as a once-per-week intravenous infusion of 90 mg/m2 over approximately 1 hour on days 1, 8, and 15 of each 28-day treatment cycle. Capivasertib 400 mg or placebo was administered orally twice per day on an intermittent weekly dosing schedule, with treatment on days 2 to 5 of weeks 1, 2, and 3 within each 28-day cycle. All treatments were continued until disease progression, development of unacceptable toxicity, or withdrawal of consent. If paclitaxel treatment was discontinued before disease progression, patients could continue to receive capivasertib or placebo alone. In case of adverse events (AEs), capivasertib or placebo could be reduced to 320 mg twice per day and subsequently to 240 mg twice per day. Capivasertib or placebo could be interrupted for up to 4 weeks for toxicity.

Tumor assessments included computed tomography scanning or magnetic resonance imaging of the chest, abdomen, and pelvis at baseline, every 8 weeks during treatment, and at progression. Patients who discontinued treatment for any reason other than progression were required to follow the same schedule of assessments until progression, initiation of another treatment, death, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to admission to this study
2. Women, age > 18 years
3. Histologically confirmed breast cancer
4. Metastatic or locally recurrent disease; locally recurrent disease must not be amenable to resection with curative intent (patients who are considered suitable for surgical or ablative techniques following potential down-staging with study treatment are not eligible)
5. Patient must have

   * At least one lesion, not previously irradiated, that can be measured accurately at baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥15mm) with CT, or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements, OR
   * lytic or mixed bone lesions in the absence of measurable disease as defined above; patients with sclerotic/osteoblastic bone lesions only in the absence of measurable disease are not eligible.
6. Radiological or clinical evidence of recurrence or progression
7. Triple-negative disease
8. Formalin fixed paraffin embedded tumour sample from the primary or recurrent cancer must be available for central testing
9. Patients must be able to swallow and retain oral medication
10. Haematologic and biochemical indices within protocol specified ranges
11. ECOG performance status 0-2
12. Non-childbearing potential. If patient is of childbearing potential, she must have a negative serum pregnancy test and agree to use adequate contraception
13. Willing and able to provide written informed consent

Exclusion Criteria:

1. Patients with confirm brain metastases or a history of primary central nervous system tumours or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases.
2. Prior chemotherapy for metastatic breast cancer
3. Radiotherapy with a wide field of radiation within 4 weeks before the first dose of study medication
4. Prior treatment with PI3K inhibitors, AKT inhibitors or mTOR inhibitors
5. Prior treatment with paclitaxel or docetaxel in the (neo)adjuvant setting within 12 months from inclusion into this study
6. Pre-existing sensory or motor polyneuropathy ≥ Grade 2 according to CTCAE
7. Malabsorption syndrome or other condition that would interfere with enteral absorption
8. Clinically significant pulmonary dysfunction
9. Prolongation defined as a QTc interval >470msecs or other significant abnormalities in rhythm, conduction or morphology of resting ECG including 2nd degree (Type II) or 3rd degree AV block or bradycardia (ventricular rate <50 beats/min)
10. Any factors that increase risk of QTc prolongation or risk of arrythmic events
11. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure NYHA Grade ≥2, or cardiac ejection fraction outside institutional range of normal or <50%
12. Clinically significant abnormalities of glucose metabolism
13. Patients with proteinuria or creatine >1.5xULN concurrent with creatinine clearance <50mL/min
14. Exposure to potent inhibitors or inducers or substrates of CYP3A4 or substrates of CYP2D6 within 2 weeks before the first dose of study treatment
15. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to study entry
16. Psychological, familial, sociological or geographical conditions that do not permit compliance with the study protocol.
17. Detained persons or prisoners
18. Pregnant or nursing women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-05-14 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Date of randomisation to date of first tumour progression or death (this can range on average between 3 weeks and 32 weeks).
  Progression-free survival, defined as the time from the date of randomisation to the date of first documented tumour progression (using RECIST 1.1) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Study Chair — Queen Mary University London; Nicholas Turner, Principal Investigator — Royal Marsden Hospital NHS- Institute of Cancer Research
Locations (46):
- France (3):
  - ICO René Gauducheau, Nantes
  - Centre André-lacassagne, Nice
  - Centre Hospitalier Prive Saint-Gregoire, Saint-Grégoire
- Institute of Clinical Oncology, Tbilisi, Georgia
- Hungary (3):
  - Országos Onkológiai Intézet, Budapest
  - University of Pécs - Clinical Center Institute of Oncotherapy, Pécs
  - Zala County Hospital Szent Rafael, Zalaegerszeg
- Romania (3):
  - Prof. Dr. I. Chiricuta Oncology Institute, Cluj-Napoca
  - Sf. Nectarie SRL Oncologie Medical Center, Craiova
  - Center of Oncology Euroclinic, Iași
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Goyang-si
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Centre, Seoul
  - Yonsei University Health System, Seoul
- United Kingdom (30):
  - Betsi Cadwaladr University Health Board, Bangor
  - Belfast Health and Social Care Trust, Belfast
  - Glan Clwyd Hospital BCU Health Board NHS Wales, Bodelwyddan
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Velindre Cancer Centre, Cardiff
  - University Hospitals Coventry and Warwickshire NHs Trust, Coventry
  - NHS Lothian, Edinburgh
  - Medway NHS Foundation Trust, Gillingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Teaching Hospitals NHs Trust, Leeds
  - Barts Health NHS Trust, London
  - University College London Hospitals, London
  - Barking, Havering and Redbridge University Hospitals NHS Trust, London
  - Guys and St Thomas' NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - Royal Marsden NHS Foundation Trust-Fulham, London
  - Imperial College Healthcare NHS Trust, London
  - Maidstone and Tunbridge Wells NHS Trust, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Southampton University Hospitals NHS Trust, Southampton
  - Southend University Hospital NHS Foundation Trust, Southend
  - University Hospital of North Staffordshire NHS Trust, Stoke-on-Trent
  - Royal Marsden - Sutton, Sutton
  - Abertawe Bro Margannwg University Health Board, Swansea
  - Royal Cornwall Hospitals NHS Trust, Truro
  - Ysbyty Wrexham Maelor Hospital, Wrexham
  - Yeovil District Hospital NHS Foundation Trust, Yeovil

REFERENCES:
- [Result] Schmid P, Abraham J, Chan S, Wheatley D, Brunt AM, Nemsadze G, Baird RD, Park YH, Hall PS, Perren T, Stein RC, Mangel L, Ferrero JM, Phillips M, Conibear J, Cortes J, Foxley A, de Bruin EC, McEwen R, Stetson D, Dougherty B, Sarker SJ, Prendergast A, McLaughlin-Callan M, Burgess M, Lawrence C, Cartwright H, Mousa K, Turner NC. Capivasertib Plus Paclitaxel Versus Placebo Plus Paclitaxel As First-Line Therapy for Metastatic Triple-Negative Breast Cancer: The PAKT Trial. J Clin Oncol. 2020 Feb 10;38(5):423-433. doi: 10.1200/JCO.19.00368. Epub 2019 Dec 16. PMID 31841354